CLINICAL TRIAL: NCT01052155
Title: Accuracy of Point of Care (POC) or In-office Urine Drug Testing (Immunoassay) in Chronic Pain Patients: A Prospective Analysis of Immunoassay and Liquid Chromatography Tandem Mass Spectometry (LC/MS/MS)
Brief Title: Accuracy of Point of Care (POC) or In-office Urine Drug Testing (Immunoassay) in Chronic Pain Patients
Status: Completed | Type: Observational
Sponsor: Pain Management Center of Paducah (Other)
Collaborators: Millennium Laboratories (Unknown)
Responsible Party: Laxmaiah Manchikanti, MD/Medical Director, Pain Management Center of Paducah and Ambulatory Surgery Center
Other Study IDs: Protocol 26
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Pain
Keywords: Controlled substances; Opioids; Benzodiazepines; Illicit drugs; Immunoassay drug testing; Point of care (POC) testing; Liquid Chromatography Tandem Mass Spectometry
MeSH Terms: conditions — Chronic Pain; Substance-Related Disorders | interventions — Immunoassay

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Urine Drug Testing — LC/MS/MS Laboratory Evaluation
  Other Names: In-office Urine Drug Testing (Immunoassay)

SUMMARY:
Accuracy of Point of Care (POC) or In-office Urine Drug Testing (Immunoassay) in Chronic Pain Patients: A Prospective Analysis of Immunoassay and Liquid Chromatography Tandem Mass Spectometry (LC/MS/MS)

DETAILED DESCRIPTION:
Recruitment is indicated in patients with chronic pain management with or without controlled substance therapy.

This is a diagnostic accuracy study performed in an interventional pain management referral center in the United States.

ELIGIBILITY:
Inclusion criteria:

• Chronic pain management with or without controlled substance therapy.

Exclusion criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain management with or without controlled substance therapy.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center, Paducah

REFERENCES:
- [Derived] Manchikanti L, Malla Y, Wargo BW, Fellows B. Comparative evaluation of the accuracy of benzodiazepine testing in chronic pain patients utilizing immunoassay with liquid chromatography tandem mass spectrometry (LC/MS/MS) of urine drug testing. Pain Physician. 2011 May-Jun;14(3):259-70. PMID 21587329
- [Derived] Manchikanti L, Malla Y, Wargo BW, Fellows B. Comparative evaluation of the accuracy of immunoassay with liquid chromatography tandem mass spectrometry (LC/MS/MS) of urine drug testing (UDT) opioids and illicit drugs in chronic pain patients. Pain Physician. 2011 Mar-Apr;14(2):175-87. PMID 21412372
- [Derived] Manchikanti L, Malla Y, Wargo BW, Cash KA, Pampati V, Damron KS, McManus CD, Brandon DE. Protocol for accuracy of point of care (POC) or in-office urine drug testing (immunoassay) in chronic pain patients: a prospective analysis of immunoassay and liquid chromatography tandem mass spectometry (LC/MS/MS). Pain Physician. 2010 Jan-Feb;13(1):E1-E22. PMID 20119473